CLINICAL TRIAL: NCT01084980
Title: A Pilot Study for Comparative Clinical Trial on the Therapeutic Effect of Tacrolimus (Prograf Cap®) in Combination With Low Dose Corticosteroid in Adult Patient With Minimal Change Nephritic Syndrome
Brief Title: Therapeutic Effect of Tacrolimus in Combination With Low Dose Corticosteroid in Adult Patient With Minimal Change Nephritic Syndrome
Acronym: MCNS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Suhnggwon Kim, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCNS001
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Minimal Change Disease
Keywords: minimal change disease; tacrolimus; corticosteroid
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Tacrolimus

ARMS (1):
- Tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — tacrolimus 0.05mg/kg bid for 12 weeks corticosteroid 0.3 - 0.5mg/kg qd
  Other Names: Prograf

SUMMARY:
The hypothesis of this study is that tacrolimus reduces the proteinuria in adult patient with minimal change nephritic syndrome.

DETAILED DESCRIPTION:
A pilot study for comparative clinical trial on the therapeutic effect of tacrolimus (Prograf cap®) in adult patient with minimal change nephritic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* from 18yrs to 80 yrs , man and women
* Minimal change disease is diagnosed by kidney biopsy
* On screening, the patient shows that the level of urine protein/creatinine ratio is over 3.0
* On screening, the patient shows that the serum albumin is below 3.0g/dL
* the patient sign on the concent form

Exclusion Criteria:

* the patient have experience to take tacrolimus or cyclosporin for 1 month
* If it is the relapse of the nephrotic syndrome, before relapse, the maintenance dose of steroid is over 0.3 mg/kg/day
* steroid dependent or steroid resistant or frequent relapse case
* uncontrolled hypertension
* pregnancy or anticipate pregnancy with 6 month
* hypersensitivity to tacrolimus or macrolide
* acute hepatitis or the level of AST or ALT is over 2 times of normal range or the level of bilirubin is over 2.0 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
remission of proteinuria | 12 weeks

SECONDARY OUTCOMES:
time to remission, relapse rate, response failure rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea